CLINICAL TRIAL: NCT04246762
Title: A Phase 1, Open-label, Study in Subjects With Rheumatoid Arthritis to Evaluate the Effect of a Single Dose of Olokizumab on the Pharmacokinetics of Substrates for CYP1A2, CYP2C9, CYP2C19, and CYP3A4
Brief Title: Study in Subjects With Rheumatoid Arthritis to Evaluate the Effect of a Single Dose of Olokizumab on the Pharmacokinetics of Substrates for CYP1A2, CYP2C9, CYP2C19 and CYP3A4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry); Thermo Fisher Scientific FS (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04041026
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate Rheumatoid Arthritis; severe Rheumatoid Arthritis; subcutaneous; Olokizumab; drug interaction; CYP450
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab; Omeprazole; Caffeine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olokizumab 128 mg +Cocktail drugs (Experimental): All subjects have received the following treatment:
  Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered with 240 mL of water on Day 1, single subcutaneous injection of Olokizumab 128 mg administered on Day 8 and second dose of Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered on Day 22
  Interventions: Drug: Olokizumab; Drug: Omeprazole; Drug: Caffeine; Drug: Warfarin+ Vitamin K; Drug: Midazolam

INTERVENTIONS:
Drug: Olokizumab — Sterile solution for subcutaneous (SC) injection, 128 mg (0.8 mL injection)
Drug: Omeprazole — Tablets, 20 mg, oral
Drug: Caffeine — Tablets, 100 mg, oral
Drug: Warfarin+ Vitamin K — Warfarin -Tablets 10 mg (containing 5 mg S-warfarin), oral. Vitamin K - solution for intravenous injection, 10 mg/mL ampoule, orally.
Drug: Midazolam — Syrup, 2 mg/mL, oral

SUMMARY:
Olokizumab (OKZ) has been shown to reverse the inhibitory effect of IL-6 on the activity of Cytochrome P450 (CYP450) isozymes CYP1A2, CYP2B6, CYP2C9, CYP2C19, and CYP3A4/5 in vitro.

The goal of the study was to assess the effect of OKZ on the pharmacokinetics (PK) of the CYP450 probe substrates, caffeine (CYP1A2), S-warfarin (CYP2C9), omeprazole (CYP2C19), and midazolam (CYP3A4) in subjects with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This was a Phase 1, open-label, 3-period, single-sequence, crossover study in subjects with RA with increased C-reactive protein (CRP).

Approximately 15 eligible subjects were planned to be enrolled at approximately 3 study centers to have at least 12 evaluable subjects completing the study. However, if necessary, additional subjects could be dosed to obtain the 12 evaluable subjects required.

There was a 35-day Screening Period, followed by a 29-day study duration: eligible patients were administered a cocktail of 4 substrates alone with following 7 days PK-sampling (Period 1); a single subcutaneous dose of 128 mg OKZ was administered (Period 2) approximately 2 weeks prior to the second administration of the cocktail with following 7-days PK-sampling (Period 3). After completion of the Period 3 patients were followed-up for 19 weeks (133 days) for safety evaluations.

Overall duration of the study was approximately 200 days (6 and a half months).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to give voluntary informed consent and sign an Informed Consent Form (ICF)
2. Male subjects and their female partners and female subjects of childbearing potential must agree to adhere to the contraceptive requirements for the study

   Female subjects of non-childbearing potential must be:

   • Surgically sterile (i.e. bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to first dosing), or

   • Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to first dosing, with a follicle stimulating hormone level at screening of ≥40 mIU/mL.
3. Body mass index of 18 kg/m2 to 29.9 kg/m2, inclusive, and body weight of 55 kg to 110 kg, inclusive, if male, and 45 kg to 100 kg, inclusive, if female.
4. Subjects must have a diagnosis of adult onset RA classified by the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 revised classification criteria for RA (Aletaha et al, 2010) for at least 12 weeks prior to Screening. If the subject was previously diagnosed according to ACR 1987 criteria, the Investigator may classify the subject per ACR 2010 retrospectively, based on medical history, and using available source data.
5. Subjects must have received Methotrexate (MTX), sulfasalazine, or hydroxychloroquine for at least 12 weeks prior to Day 1 and in stable dose for at least 6 weeks prior to Day 1 without significant Adverse events (AEs). Stable doses of MTX should be 10 mg to 25 mg weekly with folic acid (at least 5 mg weekly or equivalent). No significant side effects based on the Investigator's judgment should be observed during treatment by these agents. The maximum allowed doses of sulfasalazine and hydroxychloroquine are:

   1. Sulfasalazine: 3 g per day
   2. Hydroxychloroquine: 400 mg per day

   Note: The doses should remain stable and not be changed from the time of signing the ICF until the end of the treatment period (EOT, Day 29).
6. Subjects must have an increased CRP at Screening (of ≥1.2 × ULN).
7. Female subjects of childbearing potential must have negative pregnancy test at Screening and throughout the study until the end of study (EOS) (Day 161).

Exclusion Criteria:

1. Diagnosis of any other inflammatory arthritis or systemic inflammatory disease (e.g., gout, psoriatic or reactive arthritis, Crohn's disease, Lyme disease, juvenile idiopathic arthritis, or systemic lupus erythematosus). Osteoarthritis is classified as a degenerative disease rather than an inflammatory disease.
2. Subjects with Steinbrocker Class III or IV functional capacity (incapacitated, largely, or wholly bed ridden, or confined to a wheelchair, with little, or no self-care).
3. Prior exposure to any licensed or investigational compound directly or indirectly targeting IL-6 or IL-6R within 12 months of Day 1.
4. Treatment with DMARDs other than MTX, hydroxychloroquine, or sulfasalazine. Treatment with the following DMARDs are not allowed within the specified time period prior to Day 1:

   1. 4 weeks for azathioprine, cyclosporine, chloroquine, gold, penicillamine, minocycline, or doxycycline.
   2. 12 weeks for leflunomide unless the subject has completed the following elimination procedure at least 4 weeks prior to Day 1: Cholestyramine at a dosage of 8 grams 3 times daily for at least 24 hours or activated charcoal at a dosage of 50 grams 4 times a day for at least 24 hours.
   3. 24 weeks for cyclophosphamide.
5. Treatment with any cell-depleting therapies including anti-cluster of differentiation (CD)20 or investigational agents (eg, CAMPATH®, anti-CD4, anti-CD5, anti-CD3, and anti-CD19) with the exception of rituximab. Treatment with rituximab is not allowed within 6 months of Day 1.
6. Treatment with Tumor necrosis factor alpha inhibitor (TNFi) (including investigational proposed or licensed biosimilars) or any other biologic therapy for the treatment of RA within 12 weeks of Day 1.
7. Use of parenteral or intra-articular glucocorticoids within 4 weeks prior to Day 1.
8. Use of oral glucocorticoids greater than 10 mg/day prednisone (or equivalent) or change in dosage within 4 weeks prior to Day 1.
9. Use of indomethacin and ketorolac; other nonsteroidal anti-inflammatory drugs (NSAIDs) (with the exception of aspirin, see below) must be taken at a stable dose and route of administration for at least 2 weeks prior to Day 1.
10. Female subjects of nonchildbearing potential taking hormone replacement therapy within 4 weeks prior to Day 1.
11. Vaccination with live vaccines in the 6 weeks prior to Day 1 or planned vaccination with live vaccines during the study.
12. Participation in any other investigational drug study within 30 days or 5 times the t1/2 of the investigational drug, whichever is longer, prior to Day 1.
13. Use of aspirin or other antiplatelet agents and anticoagulants including warfarin in the 4 weeks prior to Day 1.
14. Has received any prescription or nonprescription drugs or other products (eg, herbal preparations, food products) known to be inhibitors/inducers of CYP3A4, CYP2C9, CYP2C19, or CYP1A2 within 4 weeks prior to Day 1 and for the duration of the study up to the EOT (Day 29) Visit. The use of MTX, as described in inclusion criterion #5, is permitted.
15. Use of any herbal preparations (including foods or beverages containing herbal preparations), dietary supplements, or natural medications within 14 days of Day 1.
16. Has received midazolam and/or omeprazole (or esomeprazole) within 14 days of Day 1.
17. Excessive intake of caffeine (more than 5 cups of coffee or equivalent per day) and the inability to abstain from caffeine-containing drinks and foods from 2 days prior to each cocktail administration and while inpatient (Day -1 to Day 2 and Day 21 to Day 23, respectively).
18. Poor metabolizers of CYP2C9 (genotype *2/*2, *2/*3, *3/*3) or CYP2C19 (genotype *2/*2, *2/*3, *3/*3), ultra-rapid metabolizers of CYP2C19 (*17/*17), or high sensitivity to warfarin (VKORCI genotype AA).
19. Previous participation (enrolled) in this study or another study of OKZ in case of receiving at least one OKZ dose.
20. Abnormal laboratory values as defined below. If, in the opinion of the Investigator, exclusionary results are due to laboratory error or a transient condition, these tests may be repeated once during Screening.

    a. Creatinine level ≥1.5 mg/dL (132 µmol/L) for females or ≥2.0 mg/dL (177 µmol/L) for males.

    b. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) level ≥1.5 × ULN.

    c. Platelets <150 × 10^9/L (<150,000/mm3).

    d. White blood cell count <3.0 × 10^9/L.

    e. Neutrophil count <2.0 × 10^9/L (<2000 mm3).

    f. Hemoglobin level ≤95 g/L.

    g. Glycosylated hemoglobin (HbA1c) level ≥8%.

    h. International normalized ratio above the ULN (Normal range: 0.80 or 0.90 to 1.20, males and females of all ages).
21. Subjects with concurrent viral hepatitis B or C infection as detected by blood tests at Screening (eg, positive for hepatitis B surface antigen (HBsAg), hepatitis B DNA (HBV DNA) or hepatitis C virus antibody (HCV Ab)).

    1. HBV DNA to be tested only in anti-hepatitis B core antigen (anti-HBc) positive subjects.
    2. Subject who is positive for hepatitis B surface antibody (anti-HBs) and total antiHBc but negative for HBsAg and HBV DNA, will be eligible upon qualified specialist (i.e. hepatologist) consultation with documented conclusion no additional risk is suspected for the subject.
    3. Subject who is positive for hepatitis B surface antibody (anti-HBs) but negative for HBsAg and total anti-HBc, will be eligible with no additional consultation.
22. Subjects with human immunodeficiency virus (HIV) infection.
23. Subjects with:

    1. Suspected or confirmed current active tuberculosis (TB) disease or a history of active TB disease.
    2. Close contact (ie, sharing the same household or other enclosed environment, such as a social gathering place, workplace or facility, for extended periods during the day) with an individual with active TB within 1.5 years prior to Screening.
    3. History of untreated latent TB infection (LTBI), regardless of QuantiFERON-TB Gold Plus interferon-gamma release assay (IGRA) result at Screening.
    4. Positive IGRA result at Screening. If indeterminate, the IGRA can be repeated once during Screening. If there is a second indeterminate result, the subject will be excluded.
24. Concurrent malignancy or a history of malignancy within the last 5 years (with the exception of successfully treated carcinoma of the cervix in situ or successfully treated basal cell carcinoma or squamous cell carcinoma not less than 1 year prior to Screening [and no more than 3 excised nonmelanoma skin cancers within the last 5 years prior to Screening]).
25. Subjects with a history of major bleeding, bleeding tendencies (such as any prior gastrointestinal bleeding and recent ulceration of gastrointestinal track, congenital and acquired disorders by hemostasis), or other clinically significant predisposition to bleeding according to the physician's judgment.
26. Subjects with a history or presence of severe cardiovascular conditions such as stroke, transient ischemic attack, or myocardial infarction in medical history.
27. Uncompensated congestive heart failure, or Class III or IV heart failure defined by the New York Heart Association classification.
28. Untreated, uncontrolled, or resistant arterial hypertension Grade 2 to 3 (systolic blood pressure (BP) >160 mm Hg and/or diastolic BP >100 mm Hg, based on the mean of 3 readings). If hypertension is not controlled, subjects should be excluded, and not allowed for rescreening.
29. Uncontrolled diabetes mellitus (based on the Investigator's judgment).
30. Subjects with a history or presence of any other cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, dermatological, neurological, psychiatric, hematological, or immunologic/immunodeficiency disorder(s) or any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, contraindicate subject participation in the clinical study, or clinically significant enough in the opinion of the Investigator to alter the disposition of the study treatment, or constitute a possible confounding factor for assessment of safety of the study treatment..
31. Subjects with gastrointestinal (GI) resection (eg, partial or total gastrectomy) likely to interfere with absorption of study treatment.
32. Subjects with any infection requiring any anti-infective therapy (eg, antibiotic, antiviral, or antifungal therapy) in the 4 weeks prior to Day 1, or serious or recurrent infection with history of hospitalization in the 6 months prior to Day 1 or active infection at Day 1.
33. Subjects with evidence of disseminated herpes zoster infection, zoster encephalitis, meningitis, or other nonself-limited herpes zoster infections in the 6 months prior to Day 1.
34. Subjects with planned surgery during the study (up to and including the EOT Visit,[Day 29]) or surgery ≤4 weeks prior to Screening and from which the subject has not fully recovered, as judged by the Investigator.
35. Subjects with diverticulitis or other symptomatic GI conditions that might predispose the subject to perforations, including subjects with a history of such predisposing conditions (eg, diverticulitis, GI perforation, or ulcerative colitis).
36. History of chronic alcohol or drug abuse or consumption of more than 21 units (male subjects) or 14 units (female subjects) of alcohol a week (unit = 1 glass of wine [125 mL] = 1 measure of spirits = ½ pint of beer) as judged by the Investigator.
37. Current smokers or those who have smoked or used nicotine products within the previous 3 months prior to Screening.
38. Subjects with a known hypersensitivity or contraindication to any component of the cocktail drugs or OKZ.
39. History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
40. Any self-reported symptoms of influenza-like or COVID-19 like illness in the 14 days preceding Screening OR Day 1 as per the Investigators assessment. Symptoms related to COVID-19 include, but are not limited to:

    a. Respiratory symptoms (eg, sore throat, nasal congestion, post-nasal discharge, wheezing, cough, dyspnea, and bronchial breath sounds);

    b. Non-respiratory symptoms, such as gastrointestinal symptoms (eg, nausea, vomiting, and diarrhea), neurologic symptoms (eg, anosmia, ageusia, headache), myalgia or fatigue.
41. Active SARS-CoV-2 infection as confirmed by reverse transcription polymerase chain reaction (RT-PCR) or/and positive serology at Screening.
42. Known exposure to an individual with confirmed COVID-19 or SARS-CoV-2 infection within 2 weeks before Screening OR Day 1.
43. History of COVID-19 infection in the previous 3 months before Day 1 or with sever or critical illness ever.

Note: The subject can be enrolled if all of the following criteria are fulfill:

1. had non-sever or non-critical COVID-19 infection more than 3 months before Day 1;
2. fully recovered as per official medical records which should be documented as a source document (mild sequelae of the previous infection such as dry cough, weakness should be resolved by the time of Screening);
3. there are no any concerns that the subject is infections to others;
4. there are no any other local guidelines/requirements with regards of this group of subjects.

44. Those subjects who have been at high risk of exposure before Screening, including but not limited to: Close contacts of confirmed COVID-19 cases, anyone who had to self-isolate as a result of a symptomatic household member, frontline healthcare professionals working in accident and emergency (A&E), ICU and other higher risk areas.

45. Individuals currently working with high risk of exposure to SARS-CoV-2 (eg, active healthcare workers or emergency response personnel having direct interactions with or providing direct care to patients).

46. Pregnancy and breastfeeding.

47. Other medical or psychiatric conditions or laboratory abnormalities that may increase potential risk associated with study participation and administration of study treatment, or that may affect study results interpretation and, as per the Investigator's judgment.

48. Subject's unwillingness or inability to follow the procedures outlined in the protocol.

49. Employees or relatives of the Sponsor, Contract Research Organization, or the study center personnel.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (2):
- Comac Medical Ltd, Sofia, Bulgaria
- ICS ARENSIA Exploratory Medicine SRL, a daughter company of ARENSIA Exploratory Medicine GmbH,Republican Clinical Hospital, Chisinau, Moldova

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 2 sites in 2 countries (Bulgaria and Moldova). A total of 17 subjects were enrolled into Period 1 of the study and 16 subjects each were enrolled into Period 2 and Period 3 of the study. All 17 subjects who received the first dose were enrolled into Safety Analysis Set and 16 subjects were enrolled into Pharmacokinetics (PK) and Pharmacodynamics (PD) Analysis Sets.
Groups:
- Olokizumab 128 mg + Cocktail Drugs: All subjects have received the following treatment:
  Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered with 240 mL of water on Day 1 (Period 1), single subcutaneous injection of Olokizumab 128 mg administered on Day 8 (Period 2) and second dose of Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered on Day 22 (Period 3).
  Olokizumab: Sterile solution for subcutaneous (SC) injection, 128 mg (0.8 mL injection); Omeprazole: Tablets, 20 mg, oral; Caffeine: Tablets, 100 mg, oral; Warfarin + Vitamin K: Warfarin -Tablets 10 mg (containing 5 mg S-warfarin), oral; Vitamin K - solution for intravenous injection, 10 mg/mL ampoule (orally); Midazolam: Syrup, 2 mg/mL, oral.
Period: Period 1: Cocktail Alone
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Started | 17
Completed | 16
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Period 2: Olokizumab Administration
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Started | 16
Completed | 16
Not Completed | 0
Period: Period 3: Olokizumab + Cocktail
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Started | 16
Completed | 16
Not Completed | 0
Period: Safety Follow-up
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [27 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 27.58 [23.8 to 29.8]
C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 21.996 (33.0943)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUC(0-inf)) for Caffeine, Omeprazole and Midazolam
Description: Area under the AUC from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation.
  In case of anomalous predose concentration of greater than 5% of Cmax was indicated, the PK parameters for the affected analyte and given subject were excluded from the analyses.
  Since caffeine is contained in the plethora of foods and beverages, most subjects had predose caffeine concentrations on Day 1 and Day 22 that exceeded 5% of their Maximum plasma concentration (Cmax). Caffeine PK parameter calculations and analyses were performed using concentrations adjusted by subtracting the contribution of the predose caffeine levels at each postdose timepoint using the following equation: Concentration (adjusted) = Concentration (observed) - [C predose * exp(-k*t)], with 'k' representing the patient-specific elimination rate constant (λz) determined using observed caffeine concentration data on Day 1 and Day 22 and 't' representing the actual time postdose.
Time Frame: Day 1: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24 (Day 2), 30 (Day 2, only caffeine) hours post-dose; Day 22: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24 (Day 23), 30 (Day 23, only caffeine) hours post-dose
Population: These subjects were excluded:
  For 1 subject the Percentage of AUC(0-inf) obtained by extrapolation (%AUCex) was > 20.0 % for midazolam on Day 1.
  1 subject had a quantifiable predose concentration of Omeprazole on Day 1 that exceeded 5% of Cmax.
  For 3 subjects the %AUCex exceeded 20.0 % for baseline-adjusted caffeine on Day 22 and for 1 subject - on Day 1 also. For 1 subject λz calculated from the observed caffeine concentration data on Day 1 was not adequate for baseline adjustment purposes.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
h*ng/mL
  Midazolam: number analyzed (Participants) | 15
  Midazolam | 38.23 [30.32 to 48.21]
  Midazolam + OKZ | 26.94 [21.43 to 33.86]
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 1408 [933.5 to 2124]
  Omeprazole + OKZ | 955.8 [635.3 to 1438]
  Caffeine (baseline-adjusted): number analyzed (Participants) | 14
  Caffeine (baseline-adjusted) | 21820 [17610 to 27040]
  Caffeine + OKZ (baseline-adjusted): number analyzed (Participants) | 13
  Caffeine + OKZ (baseline-adjusted) | 26830 [21580 to 33340]
Statistical Analysis 1: Comparison: Olokizumab 128 mg + Cocktail Drugs; Estimate of the mean difference between treatments (midazolam (as part of a 4-drug oral cocktail) after OKZ administration compared to midazolam (as part of a 4-drug oral cocktail) administrated alone) and its corresponding 90% confidence interval (CI) were calculated. The mean difference and the CI were back transformed to the original scale to obtain estimates of the geometric mean ratio and the associated 90% CI; Test type: Other; geometric LS mean ratio of AUC (0-inf)) = 70.46, 90% CI 2-sided [60.62 to 81.91] — Results based on a linear mixed model for the log-transformed values of PK parameters of midazolam with a fixed effect for treatment and a random effect for subject
Statistical Analysis 2: Comparison: Olokizumab 128 mg + Cocktail Drugs; Estimate of the mean difference between treatments (omeprazole (as part of a 4-drug oral cocktail) after OKZ administration compared to omeprazole (as part of a 4-drug oral cocktail) administrated alone) and its corresponding 90% confidence interval (CI) were calculated. The mean difference and the CI were back transformed to the original scale to obtain estimates of the geometric mean ratio and the associated 90% CI; Test type: Other; geometric LS mean ratio of AUC (0-inf)) = 67.87, 90% CI 2-sided [56.73 to 81.21] — Results based on a linear mixed model for the log-transformed values of PK parameters of omeprazole with a fixed effect for treatment and a random effect for subject
Statistical Analysis 3: Comparison: Olokizumab 128 mg + Cocktail Drugs; Estimate of the mean difference between treatments (caffeine (as part of a 4-drug oral cocktail) after OKZ administration compared to caffeine (as part of a 4-drug oral cocktail) administrated alone) and its corresponding 90% confidence interval (CI) were calculated. The mean difference and the CI were back transformed to the original scale to obtain estimates of the geometric mean ratio and the associated 90% CI; Test type: Other; geometric LS mean ratio of AUC (0-inf)) = 122.92, 90% CI 2-sided [107.98 to 139.93] — Results based on a linear mixed model for the log-transformed values of baseline-adjusted PK parameters of caffeine with a with fixed effect for treatment and a random effect for subject

2. Primary Outcome: AUC From Time Zero to the Time "t" (AUC(0-last)) for S-warfarin
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration, calculated by linear up/log down trapezoidal summation for S-warfarin (10 mg warfarin contains 5 mg S-warfarin)
Time Frame: Day 1: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24(Day 2), 48(Day 3), 72 (Day 4), 120 (Day 6), 168 (Day 8) hours post-dose; Day 22: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24(Day 23), 48(Day 24), 72 (Day 25), 120 (Day 27), 168 (Day 29) hours post-dose
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Groups:
- Olokizumab 128 mg + Cocktail Drugs: All subjects have received the following treatment:
  Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered with 240 mL of water on Day 1 (Period 1), single subcutaneous injection of Olokizumab 128 mg administered on Day 8 (Period 2) and second dose of Cocktail drugs (Omeprazole + Caffeine + Warfarin (+ vitamin K solution) + Midazolam) orally administered on Day 22 (Period 3).
  Olokizumab: Sterile solution for subcutaneous (SC) injection, 128 mg (0.8 mL injection); Omeprazole: Tablets, 20 mg, oral; Caffeine: Tablets, 100 mg, oral; Warfarin + Vitamin K: Warfarin - Tablets 10 mg (containing 5 mg S-warfarin), oral; Vitamin K - solution for intravenous injection, 10 mg/mL ampoule (orally); Midazolam: Syrup, 2 mg/mL, oral.
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
h*ng/mL
  S-Warfarin | 21350 [18360 to 24820]
  S-Warfarin + OKZ | 19390 [16680 to 22540]
Statistical Analysis 1: Comparison: Olokizumab 128 mg + Cocktail Drugs; Estimate of the mean difference between treatments (S-warfarin (as part of a 4-drug oral cocktail) after OKZ administration compared to initial S-warfarin administrated alone (as part of a 4-drug oral cocktail)) and its corresponding 90% confidence interval (CI) was calculated. The mean difference and the CI were back transformed to the original scale to obtain estimate of the geometric mean ratio and the associated 90% CI; Test type: Other; geometric LS mean ratio of AUC (0-last)) = 90.83, 90% CI 2-sided [86.72 to 95.13] — Results based on a linear mixed model for the log-transformed values of PK parameters of S-warfarin with a fixed effect for treatment and a random effect for subject

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for All Cocktail Substrates
Description: Cmax for all cocktail substrates (caffeine, omeprazole, midazolam and S-warfarin), obtained directly from the observed concentration versus time data.
  In case of anomalous predose concentration of greater than 5% of Cmax was indicated, the PK parameters for the affected analyte and given subject were excluded from the analyses.
  Since caffeine is contained in the plethora of foods and beverages, most subjects had predose caffeine concentrations on Day 1 and Day 22 that exceeded 5% of their Cmax. Caffeine PK parameter calculations and analyses were performed using concentrations adjusted by subtracting the contribution of the predose caffeine levels at each postdose timepoint using the following equation: Concentration (adjusted) = Concentration (observed) - [C predose * exp(-k*t)], with 'k' representing the patient-specific elimination rate constant (λz) determined using observed caffeine concentration data on Day 1 and Day 22 and 't' representing the actual time postdose.
Time Frame: Day 1: pre-dose, 0.5 - 24, 30 (only caffeine), 48 (only S-warfarin), 72 (only S-warfarin), 120 (only S-warfarin), 168 (only S-warfarin) hours post-dose; Day 22: pre-dose, 0.5 - 24, 30 (only caffeine), 48 - 168 (only S-warfarin) hours post-dose
Population: One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax and all PK parameters were excluded from summary presentations and statistical analysis for that study day.
  For one subject lambda-z (observed) of caffeine was not adequate for baseline adjustment and Cmax was excluded from summary presentations and statistical analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
ng/mL
  Midazolam | 13.29 [11.08 to 15.93]
  Midazolam + OKZ | 9.101 [7.593 to 10.91]
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 668.6 [522.4 to 855.6]
  Omeprazole + OKZ | 491.7 [385.2 to 627.7]
  Caffeine (baseline adjusted): number analyzed (Participants) | 15
  Caffeine (baseline adjusted) | 2803 [2570 to 3057]
  Caffeine + OKZ (baseline adjusted) | 2746 [2523 to 2990]
  S-Warfarin | 627.0 [571.5 to 688.0]
  S-Warfarin + OKZ | 641.5 [584.6 to 703.9]
Statistical Analysis 1: Comparison: Olokizumab 128 mg + Cocktail Drugs; [analysis description as in outcome 1, analysis 1]; Test type: Other; geometric LS mean ratio of Cmax = 68.50, 90% CI 2-sided [59.46 to 78.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Olokizumab 128 mg + Cocktail Drugs; [analysis description as in outcome 1, analysis 2]; Test type: Other; geometric LS mean ratio of Cmax = 73.54, 90% CI 2-sided [64.18 to 84.27] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Olokizumab 128 mg + Cocktail Drugs; [analysis description as in outcome 1, analysis 3]; Test type: Other; geometric LS mean ratio of Cmax = 97.99, 90% CI 2-sided [91.36 to 105.09] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Olokizumab 128 mg + Cocktail Drugs; Estimate of the mean difference between treatments (S-warfarin (as part of a 4-drug oral cocktail) after OKZ administration compared to initial S-warfarin administrated alone (as part of a 4-drug oral cocktail)) and its corresponding 90% confidence interval (CI) was calculated. The mean difference and the CI were back transformed to the original scale to obtain estimate of the geometric mean ratio and the associated 90% CI. The sample size computation was based on results reported for sirukumab; Test type: Other; geometric LS mean ratio of Cmax = 102.30, 90% CI 2-sided [94.80 to 110.39] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Plasma AUC(0-last) for Cocktail Parent Compounds (for Caffeine, Omeprazole and Midazolam)
Description: AUC from time zero to the time of the last quantifiable concentration, calculated by linear up/log down trapezoidal summation for Caffeine, Omeprazole, Midazolam.
  In case of anomalous predose concentration of greater than 5% of Cmax was indicated, the PK parameters for the affected analyte and given subject were excluded from the analyses. Since caffeine is contained in the plethora of foods and beverages, most subjects had predose caffeine concentrations on Day 1 and Day 22 that exceeded 5% of their Cmax. Caffeine PK parameter calculations and analyses were performed using concentrations adjusted by subtracting the contribution of the predose caffeine levels at each postdose timepoint using the following equation: Concentration (adjusted) = Concentration (observed) - [C predose * exp(-k*t)], with 'k' representing the patient-specific elimination rate constant (λz) determined using observed caffeine concentration data on Day 1 and Day 22 and 't' representing the actual time postdose.
Time Frame: as for outcome 1
Population: One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax and all PK parameters were excluded from summary presentations and statistical analysis for that study day.
  For one subject lambda-z (observed) of caffeine was not adequate for baseline adjustment and AUC(0-last) was excluded from summary presentations and statistical analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
h*ng/mL
  Midazolam | 36.77 (43.0)
  Midazolam + OKZ | 24.73 (49.6)
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 1461 (92.2)
  Omeprazole + OKZ | 951.1 (86.3)
  Caffeine (baseline-adjusted): number analyzed (Participants) | 15
  Caffeine (baseline-adjusted) | 21860 (42.2)
  Caffeine (baseline-adjusted) + OKZ | 26910 (42.8)

5. Secondary Outcome: Plasma AUC From Time Zero to Infinity (AUC(0-inf)) for Cocktail Parent Compounds (for S-warfarin)
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation for S-warfarin (10 mg warfarin contains 5 mg S-warfarin).
Time Frame: Day 1: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24, 48, 72, 120, 168 hours post-dose; Day 22: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 7, 12, 24, 48, 72, 120, 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
h*ng/mL
  S-warfarin | 21350 (29.4)
  S-warfarin + OKZ | 19390 (28.7)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Cocktail Parent Compounds
Description: tmax for cocktail parent compounds (caffeine, S-warfarin, omeprazole and midazolam), obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 3
Population: One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax and all PK parameters were excluded from summary presentations and statistical analysis for that study day.
  For one subject lambda-z (observed) of caffeine was not adequate for baseline adjustment and tmax was excluded from summary presentations and statistical analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
hours
  Midazolam | 0.500 [0.48 to 1.03]
  Midazolam + OKZ | 0.533 [0.50 to 1.03]
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 2.000 [1.00 to 3.03]
  Omeprazole + OKZ | 2.000 [1.00 to 4.03]
  Caffeine (baseline-adjusted): number analyzed (Participants) | 15
  Caffeine (baseline-adjusted) | 0.533 [0.23 to 2.00]
  Caffeine (baseline-adjusted) + OKZ | 0.558 [0.50 to 2.03]
  S-Warfarin | 1.500 [0.50 to 3.03]
  S-Warfarin + OKZ | 1.500 [0.25 to 4.00]

7. Secondary Outcome: Terminal Half-life (t1/2) for Cocktail Parent Compounds
Description: Terminal half-life (t1/2) for cocktail parent compounds (caffeine, S-warfarin (10 mg warfarin contains 5 mg S-warfarin), omeprazole, and midazolam)
Time Frame: Day 1: pre-dose, 0.5 - 24, 30 (only caffeine), 48 - 168 (only S-warfarin) hours post-dose; Day 22: pre-dose, 0.5 - 24, 30 (only caffeine), 48 - 168 (only S-warfarin) hours post-dose
Population: One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax and all PK parameters were excluded from summary presentations and statistical analysis for that study day.
  For one subject lambda-z (observed) of caffeine was not adequate for baseline adjustment and t1/2 was excluded from summary presentations and statistical analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
hours
  Midazolam | 6.726 (28.6)
  Midazolam + OKZ | 6.520 (32.8)
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 1.279 (59.8)
  Omeprazole + OKZ | 0.9859 (51.5)
  Caffeine (baseline-adjusted): number analyzed (Participants) | 15
  Caffeine (baseline-adjusted) | 6.375 (43.1)
  Caffeine (baseline-adjusted) + OKZ | 8.046 (48.2)
  S-Warfarin | 43.94 (13.6)
  S-Warfarin + OKZ | 38.57 (14.6)

8. Secondary Outcome: Elimination Rate Constant (λz) for Cocktail Parent Compounds
Description: elimination rate constant (λz) for cocktail parent compounds (caffeine, S-warfarin (10 mg warfarin contains 5 mg S-warfarin), omeprazole, and midazolam), determined by linear regression of the terminal points of the log-linear concentration-time curve. The Best Fit method utilized by WinNonlin was used to identify the terminal linear phase of the concentration-time profile, with visual assessment and adjustment of the selected data points by the PK scientist if warranted.
Time Frame: as for outcome 7
Population: One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax and all PK parameters were excluded from summary presentations and statistical analysis for that study day.
  For one subject lambda-z (observed) of caffeine was not adequate for baseline adjustment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hours
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
1/hours
  Midazolam | 0.1031 (28.6)
  Midazolam + OKZ | 0.1063 (32.8)
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 0.5418 (59.8)
  Omeprazole + OKZ | 0.7031 (51.5)
  Caffeine (baseline-adjusted): number analyzed (Participants) | 15
  Caffeine (baseline-adjusted) | 0.1087 (43.1)
  Caffeine (baseline-adjusted) + OKZ | 0.08615 (48.2)
  S-Warfarin | 0.01578 (13.6)
  S-Warfarin + OKZ | 0.01797 (14.6)

9. Secondary Outcome: Apparent Systemic Clearance (CL/F) for Cocktail Parent Compounds
Description: Apparent systemic clearance (CL/F) for cocktail parent compounds (caffeine, omeprazole, and midazolam), calculated as dose divided by AUC(0-inf).
  In case of anomalous predose concentration of greater than 5% of Cmax was indicated, the PK parameters for the affected analyte and given subject were excluded from the analyses. Since caffeine is contained in the plethora of foods and beverages, most subjects had predose caffeine concentrations on Day 1 and Day 22 that exceeded 5% of their Cmax. Caffeine PK parameter calculations and analyses were performed using concentrations adjusted by subtracting the contribution of the predose caffeine levels at each postdose timepoint using the following equation: Concentration (adjusted) = Concentration (observed) - [C predose * exp(-k*t)], with 'k' representing the patient-specific elimination rate constant (λz) determined using observed caffeine concentration data on Day 1 and Day 22 and 't' representing the actual time postdose.
Time Frame: as for outcome 7
Population: These subjects were excluded:
  For one subject the %AUCex was > 20.0% for midazolam on Day 1. For 3 subjects the %AUCex exceeded 20.0 % for baseline-adjusted caffeine on Day 22 and for 1 subject - on Day 1 also. For 1 subject λz calculated from the observed caffeine concentration data on Day 1 was not adequate for baseline adjustment purposes.
  One subject had a quantifiable predose concentration of omeprazole on Day 1 that exceeded 5% of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hours
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
L/hours
  Midazolam: number analyzed (Participants) | 15
  Midazolam | 53.23 (41.4)
  Midazolam + OKZ | 74.24 (50.2)
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 13.58 (94.3)
  Omeprazole + OKZ | 20.93 (86.9)
  Caffeine (baseline-adjusted): number analyzed (Participants) | 14
  Caffeine (baseline-adjusted) | 4.582 (37.9)
  Caffeine (baseline-adjusted) + OKZ: number analyzed (Participants) | 13
  Caffeine (baseline-adjusted) + OKZ | 3.805 (40.9)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Cocktail Parent Compounds
Description: Vz/F during terminal phase for cocktail parent compounds (caffeine, omeprazole and midazolam), calculated as dose divided by [λz *AUC(0-inf)] In case of anomalous predose concentration of greater than 5% of Cmax was indicated, the PK parameters for the affected analyte and given subject were excluded from the analyses. Since caffeine is contained in the plethora of foods and beverages, most subjects had predose caffeine concentrations on Day 1 and Day 22 that exceeded 5% of their Cmax. Caffeine PK parameter calculations and analyses were performed using concentrations adjusted by subtracting the contribution of the predose caffeine levels at each postdose timepoint using the following equation: Concentration (adjusted) = Concentration (observed) - [C predose * exp(-k*t)], with 'k' representing the patient-specific elimination rate constant (λz) determined using observed caffeine concentration data on Day 1 and Day 22 and 't' representing the actual time postdose.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
L
  Midazolam: number analyzed (Participants) | 15
  Midazolam | 492.6 (35.4)
  Midazolam + OKZ | 698.3 (43.3)
  Omeprazole: number analyzed (Participants) | 15
  Omeprazole | 25.06 (31.4)
  Omeprazole + OKZ | 29.76 (33.4)
  Caffeine (baseline-adjusted): number analyzed (Participants) | 14
  Caffeine (baseline-adjusted) | 38.86 (19.9)
  Caffeine (baseline-adjusted) + OKZ: number analyzed (Participants) | 13
  Caffeine (baseline-adjusted) + OKZ | 37.70 (37.70)

11. Secondary Outcome: Plasma Concentrations (Cmax) for Olokizumab
Description: Maximum concentration obtained directly from the observed concentration versus time data for Olokizumab.
Time Frame: Predose: within 30 min of OKZ administration on Day 8; postdose: Day 9, Day 15 (sample collection clock-matched to Day 8 sample), Day 22 (collected prior to administration of DDI cocktail), Day 24, Day 29 (sample collection clock-matched to Day 22 sample)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
ng/mL | 15670 [5030 to 24100]

12. Secondary Outcome: Change in Interleukin-6 (IL-6) Concentrations Collected Periodically Throughout the Study
Description: Blood sampling for the measurement of IL-6 were performed at Screening, prior to dosing with the cocktail on Day 1, prior to dose administration with OKZ on Day 8, and post OKZ dose administration on Day 9, Day 15, Day 22 (prior to dose administration of the cocktail on Day 22), and Day 29, which were considered the EOT visit.
Time Frame: Days 1, 8, 9, 15, 22, 29
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
pg/mL
  Baseline | 26.224 (35.0576)
  Day 8 | 16.414 (20.2591)
  Change from Baseline on Day 8 | -9.810 (34.8049)
  Day 9 | 2.518 (1.2827)
  Change from Baseline on Day 9 | -23.706 (35.4123)
  Day 15 | 6.434 (6.7420)
  Change from Baseline on Day 15 | -19.790 (35.0774)
  Day 22 | 6.796 (7.5603)
  Change from Baseline on Day 22 | -19.429 (35.4360)
  Day 29 | 5.699 (4.8192)
  Change from Baseline on Day 29 | -20.526 (34.8727)

13. Secondary Outcome: Change in C-reactive Protein (CRP) Concentrations Collected Periodically Throughout the Study
Description: Blood sampling for the measurement of CRP were performed at Screening, prior to dosing with the cocktail on Day 1, prior to dose administration with OKZ on Day 8, and post OKZ dose administration on Day 9, Day 15, Day 22 (prior to dose administration of the cocktail on Day 22), and Day 29, which were considered the EOT visit.
Time Frame: Days 1, 8, 9, 15, 22, 29
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
Number analyzed (Participants) | 16
mg/L
  Baseline | 22.969 (33.9274)
  Day 8 | 15.153 (15.3990)
  Change from Baseline on Day 8 | -7.817 (26.8275)
  Day 9 | 11.783 (11.5188)
  Change from Baseline on Day 9 | -11.187 (29.3898)
  Day 15 | 2.266 (2.0937)
  Change from Baseline on Day 15 | -20.703 (34.3184)
  Day 22 | 2.044 (2.5411)
  Change from Baseline on Day 22 | -20.926 (34.5988)
  Day 29 | 2.312 (2.8719)
  Change from Baseline on Day 29 | -20.657 (34.8682)

ADVERSE EVENTS:
Time Frame: From the signing of the Informed Consent Form (ICF) until the final end of study (EOS) telephonic follow-up visit (Day 161 ±10 days)
Description: Safety population included all subjects who received at least 1 dose of study treatment (CYP450 probe cocktail or OKZ). Subjects were analyzed according to the treatment they received.
Arm/Group | Olokizumab 128 mg + Cocktail Drugs
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olokizumab 128 mg + Cocktail Drugs (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Blood Cholesterol Increased (Investigations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04246762/Prot_SAP_000.pdf